CLINICAL TRIAL: NCT02243254
Title: Prevention of Remifentanil-induced Postoperative Hyperalgesia With Intravenous Ibuprofen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ibuprofen_hyperalgesia
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Ibuprofen; Remifentanil; Hyperalgesia; Pain, Postoperative
MeSH Terms: conditions — Hyperalgesia; Pain, Postoperative | interventions — Remifentanil; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- high dose remifentanil without ibuprofen (Placebo Comparator): remifentanil target-controlled infusion effect-site concentration 4 ng/ml normal saline before surgical incision
  Interventions: Drug: high dose remifentanil
- low dose remifentanil without ibuprofen (Placebo Comparator): remifentanil target-controlled infusion effect-site concentration 1 ng/ml normal saline before surgical incision
  Interventions: Drug: low dose remifentanil
- high dose remifentanil with ibuprofen (Active Comparator): remifentanil target-controlled infusion effect-site concentration 4 ng/ml Intravenous ibuprofen 800 mg before surgical incision
  Interventions: Drug: high dose remifentanil; Drug: Ibuprofen
- low dose remifentanil with ibuprofen (Active Comparator): remifentanil target-controlled infusion effect-site concentration 1 ng/ml Intravenous ibuprofen 800 mg before surgical incision
  Interventions: Drug: Ibuprofen; Drug: low dose remifentanil

INTERVENTIONS:
Drug: high dose remifentanil — high dose remifentanil
  Arms: high dose remifentanil with ibuprofen; high dose remifentanil without ibuprofen
Drug: Ibuprofen — intravenous ibuprofen
  Arms: high dose remifentanil with ibuprofen; low dose remifentanil with ibuprofen
Drug: low dose remifentanil — low dose remifentanil
  Arms: low dose remifentanil with ibuprofen; low dose remifentanil without ibuprofen

SUMMARY:
Postoperative hyperalgesia has been reported after intraoperative administration of small or high-dose remifentanil. Cyclooxygenase inhibitor exhibit preventive effects on the development of opioid-induced hyperalgesia. The aim of this study is to evaluate the preventive effect of intravenous ibuprofen (Caldolor®) on remifentanil-induced hyperalgesia

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective pancreaticoduodenectomy

Exclusion Criteria:

* Patients with chronic pain
* Patients with psychiatric disease
* Patients with nonsteroidal antiinflammatory drugs allergy
* Patients with renail dysfunction
* History of drug addiction
* Pregnant patient
* Inability to use a PCA device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
cumulative morphine consumption | postoperative 48 hours
  cumulative patient-controlled analgesia (PCA) morphine consumption

SECONDARY OUTCOMES:
Pain score | postoperative 1, 3, 6,12, 24, 48 hours Pain score
  visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea